CLINICAL TRIAL: NCT01548170
Title: A Phase I, Pilot, Dose Finding Clinical Trial to Assess the Interaction Between Sunitinib and Ketoconazole to Reduce the Dose and Cost of Sunitinib for National Health System
Brief Title: To Assess the Interaction Between Sunitinib and Ketoconazole to Reduce the Dose and Cost of Sunitinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KS-ONCOFARMA-01; 2010-023739-41 (EudraCT Number)
Record Dates: First submitted 2011-12-23; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Cancer
Keywords: Pharmacokinetic; Sunitinib; Ketoconazol; interaction, Phase I
MeSH Terms: conditions — Neoplasms | interventions — Sunitinib; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Sunitinib 50mg (Active Comparator): Sunitinib 50 mg administered as a single dose.
  Interventions: Drug: Sunitinib
- Sunitinib 37.5mg + Ketoconazol 200mg (Experimental): The drugs will be administered as follows:
  * Sunitinib 37.5mg oral single dose.
  * Ketoconazole 200 mg orally, once daily for 6 days. (Combination with sunitinib will be performed on day 4)
  Interventions: Drug: Sunitiinb and Ketoconazol
- Sunitinib 37.5 mg + Ketoconazol 400 mg (Experimental): The drugs will be administered as follows:
  * Sunitinib 37.5mg oral single dose.
  * Ketoconazole 400 mg orally, once daily for 6 days. (Combination with sunitinib will be performed on day 4)
  Interventions: Drug: Sunitinib and Ketoconazol
- Sunitinib 25mg + Ketoconazol 200mg (Experimental): The drugs will be administered as follows:
  * Sunitinib 25mg oral single dose.
  * Ketoconazole 200 mg orally, once daily for 6 days. (Combination with sunitinib will be performed on day 4)
  Interventions: Drug: Sunitinib and Ketoconazol
- Sunitinib 25mg + Ketoconazol 400mg (Experimental): The drugs will be administered as follows:
  * Sunitinib 25mg oral single dose.
  * Ketoconazole 400 mg orally, once daily for 6 days. (Combination with sunitinib will be performed on day 4)
  Interventions: Drug: Sunitinib and Ketoconazol

INTERVENTIONS:
Drug: Sunitinib — One capsule of sunitinib 50 mg orally. Single dose
  Arms: Sunitinib 50mg
Drug: Sunitinib and Ketoconazol — Sunitinib capsule 37.5mg. Single dose Ketoconazol 2 tablets of 200mg administered daily during 6 days.
  Arms: Sunitinib 37.5 mg + Ketoconazol 400 mg
Drug: Sunitiinb and Ketoconazol — Sunitinib capsule 37.5mg. Single dose Ketoconazol 1 tablet of 200mg administered daily during 6 days.
  Arms: Sunitinib 37.5mg + Ketoconazol 200mg
Drug: Sunitinib and Ketoconazol — Sunitinib capsule 25mg. Single dose Ketoconazol 1 tablet of 200mg administered daily during 6 days.
  Arms: Sunitinib 25mg + Ketoconazol 200mg
Drug: Sunitinib and Ketoconazol — Sunitinib capsule 25mg. Single dose Ketoconazol 2 tablets of 200mg administered daily during 6 days.
  Arms: Sunitinib 25mg + Ketoconazol 400mg

SUMMARY:
Sunitinib is an ATP competitive tyrosine kinase inhibitor of several membrane receptors including VEGFR-1, -2, and -3, PDGFR-α and -β, c-KIT, CSF-1R, FLT-3, and RET. Through this molecular mode of action, sunitinib is able to avoid tumoral angiogenesis and proliferation. Sunitinib is already approved by the FDA, EMEA and AEMPS for the treatment of patients with metastatic renal cell carcinomas and those with metastatic gastrointestinal stromal tumors (GIST) with progression or intolerance to imatinib.

Suntinib has recently reported to be superior than placebo in terms of response rate (9.3% vs. 0%; p<0.05), progression free survival (11.4 vs. 5,5 months; HR 0.41;p<0.05), and overall survival (HR 0.40;p<0.05) when administered in a phase 3 trial to patients with advanced pancreatic neuroendocrine tumors (NETs).

Sunitinib is an expensive drug that drains the budget of health public system therefore it demands a rational drug use.

Sunitinib is metabolized by CYP3A4, that belongs to the P450 cytochrome system in the liver. Most of the drug is eliminated in faeces and only 16% by urine. Sunitinib has no food-effect when taken with meals. Pharmacokinetics parameters did not differ between cancer patients and healthy volunteers.

Houk et al. Showed that the area under the curve of plasmatic concentration of sunitinib and its active metabolite did correlate with clinical outcome. In other words, the higher plasma concentration area under the curve the highest rates of radiological response, progression free and overall survival rates.

Ketoconazol is an antifungal drug that inhibits the CY3A4 inducing an elevation of peak plasma levels of other drugs administered simultaneously and that are metabolized by the same system. In the labeling sheet of sunitinib it is said that ketoconazol induced a 49% and 51% of increase of plasmatic sunitinib Cmax y AUC0-∞ when both drugs were administered together. This fact makes that the investigatorspropose that by administering both drugs simultaneously the investigators could reduce sunitinib dose by a lower metabolization with similar plasma concentration. The dose reduction would impact in drug cost.

Here the investigators propose to determine the most optimal combination dose of sunitinib (25 mg or 37.5 mg) and ketoconazol (200mg o 400mg) by which the investigators could have plasmatic bioequivalent concentrations compared with single dose of sunitinib 50mg.

Each volunteer will be assigned to a treatment arm (Arm A and Arm B). Volunteers included in Arm A will take: sunitinib 50 mg, sunitinib 37.5 mg + ketoconazole 200 mg and sunitinib 37.5 mg + 400 mg ketoconazole. Volunteers included in Arm B will take: sunitinib 50 mg, sunitinib 25 mg + ketoconazole 200 mg and sunitinib 25 mg + 400 mg ketoconazole

DETAILED DESCRIPTION:
This is a phase I, pilot, open, randomized, parallel, and cross-over trial to assess the interaction between three different dose levels of sunitinib (50 mg, 37.5 mg, and 25 mg) and two dose levels of ketoconazole (200 mg and 400 mg) in 12 healthy volunteers (6 voluunteers in each group of treatment) Each volunteer will be assigned to a treatment arm (Arm A and Arm B. Volunteers included in Arm A will take: sunitinib 50 mg, sunitinib 37.5 mg + ketoconazole 200 mg and sunitinib 37.5 mg + 400 mg ketoconazole. Volunteers included in Arm B will take: sunitinib 50 mg, sunitinib 25 mg + ketoconazole 200 mg and sunitinib 25 mg + 400 mg ketoconazole

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals men who give their written consent to participate in the study, after having received information about the design, the project objectives, the risks and that at any moment they can refuse their cooperation.
* Age between 18 and 35 years.
* Subjects with a BMI that is between 19 and 28.
* Healthy subjects, without any organic or psychological pathology.
* Clinical history and physical examination within normal limits.
* Lack of clinically relevant abnormalities in blood test (hematology, biochemistry, virology) and urine test
* Vital signs and electrocardiographic recording in the normal range.

Exclusion Criteria:

* Subjects suffering from organic or psychological pathology. Prior to the inclusion of any volunteer it should be considered all security parameters mentioned in the protocol (biochemical markers of kidney damage and / or liver out of the normal range set by the laboratory).
* Subjects who have received prescription drug treatment in the last 15 days or any medication within 48 hours before receiving study medication.
* Known hypersensitivity to any drug
* Suspected of drug abuse

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Sunitinib pharmacokinetic parameters (Maximum plasma concentration (Cmax) and Area under the plasma concentration curve (AUC0-72) obtained in the different treatment groups. | Up to 72 hours postdose for each period
  On the fourth day of each period patient will be hospitalized in the clinical trial unit in order to obtain plasma concentrations previous to the administration of the corresponding dose and at the following times port-administration: 2h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 11h, 12h, 14h, 16h, 24h, 36h, 48h amd 72h. These measures will be calculated in order to describe the pharmacokinetic profile of each treatment arm.

SECONDARY OUTCOMES:
Other Sunitinib pharmacokinetic parameters (first time to reach Cmax (tmax) and Area under the plasma concentration curve (AUC0-Inf) obtained in the different treatment groups. | Up to 72 hours postdose for each period
  On the fourth day of each period patient will be hospitalized in the clinical trial unit in order to obtain plasma concentrations previous to the administration of the corresponding dose and at the following times port-administration: 2h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 11h, 12h, 14h, 16h, 24h, 36h, 48h amd 72h. These measures will be calculated in order to describe the pharmacokinetic profile of each treatment arm.
Coefficient of variation of AUC and Cmax | 9 months
  To estimate the actual coefficient of variation of AUC and Cmax of sunitinib in our environment when given alone and in combination with ketoconazole.
Change in QT interval | On day 4 of each period
  An ECG to measure the QT interval will be performed coinciding with blood samples taken basal and at 6h, 8h, 10h, 12h and 72 h after drug administration in each period.
Adverse events reported | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Grande Pulido, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Madrid, Spain